CLINICAL TRIAL: NCT02007291
Title: Good Rate of Clinical Response to Cholinesterase Inhibitors in Mild and Moderate Alzheimer's Disease After Three Months of Treatment
Brief Title: Good Rate of Clinical Response to Cholinesterase Inhibitors in Alzheimer's Disease After Three Months of Treatment
Acronym: NINDS-AIREN
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Luís Felipe José Ravic de Miranda, Physician, Geriatrician, MD, PhD student, Federal University of Minas Gerais
Other Study IDs: 0172 / 2010
Record Dates: First submitted 2013-08-18; First posted 2013-12-10 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Late Onset Alzheimer
Keywords: Alzheimer, MMSE, response, colinesterase inhibitors (ChEI)
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood sample was drawn from the patients on the first consultation for use in DNA extraction and Apolipoprotein E (APOE) genotyping. For the patients who were taking donepezil, after three, six and twelve months of treatment another blood sample were also drawn, separated in plasma and kept into the freezer at - 70 Celsius degree for further analysis of serum level of donepezil.
Oversight: Data Monitoring Committee: No

SUMMARY:
Life expectancy in Brazil has increased markedly over the last 30 years. Hence, age-related disorders, such as Alzheimer's disease (AD), warrant special attention due to their high prevalence in the elderly. Pharmacologic treatment of AD is based on cholinesterase inhibitors (ChEI) and memantine, leading to modest clinical benefits both in the short and long-term.

However, clinical response is heterogeneous and needs further investigation. Objective: To investigate the rate of response to ChEI in AD after three months of treatment. Methods: Patients with mild or moderate dementia due to probable AD or to AD associated with cerebrovascular disease were included in the study.

DETAILED DESCRIPTION:
The subjects were assessed at baseline and again after three months of ChEI treatment. Subjects were submitted to the Mini-Mental State Examination (MMSE), Mattis Dementia Rating Scale, Katz Basic Activities of Daily Living, Pfeffer Functional Activities Questionnaire, Neuropsychiatric Inventory and Cornell Scale for Depression in Dementia. Good response was defined by a gain of ≥2 points on the MMSE after three months of treatment in relation to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the National Institute on Aging and the Alzheimer's Association diagnostic criteria of probable AD dementia or the NINDS-AIREN (National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences) diagnostic criteria of AD with cerebrovascular disease (AD + CVD)
* Patients presenting mild or moderate dementia according to the Clinical Dementia Rating (CDR), i.e., CDR 1 or 2, respectively

Exclusion Criteria:

* Patients treated with ChEI or memantine before study entry
* Patients diagnosed with frontotemporal dementia, dementia with Lewy bodies or vascular dementia,
* Patients with CDR 3
* Illiterate patients
* Patients with different comorbidities, with signs of clinical decompensation

Ages: 59 Years to 93 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A longitudinal, naturalist study, conducted at the Geriatric Outpatient Clinic of the Hospital das Clínicas at the Federal University of Minas Gerais (UFMG), in Belo Horizonte (MG), Brazil.
  The sample comprised patients evaluated from June, 2009 until October, 2011.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2009-06; Primary Completion 2011-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Caramelli, MD, PhD, Study Chair — Federal University of Minas Gerais

RESULTS

PARTICIPANT FLOW:
Groups:
- CDR1 Patients Taking Cholinesterase Inhibitors; CDR2 Patients Taking Cholinesterase Inhibitors: The sample comprised patients evaluated from June, 2009 until October, 2011.During this period, 71 patients were evaluated at baseline and after 3 month-treatment. Donepezil, rivastigmine or galantamine were prescribed to the patients according to the clinicians' preferences. The target dosages considered for treatment effect evaluation were 5 to 10 mg for donepezil, 16 to 24 mg for galantamine and 6 to 12 mg for rivastigmine. The first investigator (LFJRM) did not have any influence on the prescription.
Period: Overall Study
Arm/Group | CDR1 Patients Taking Cholinesterase Inhibitors | CDR2 Patients Taking Cholinesterase Inhibitors
Started | 48 | 23
Completed | 48 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Taking Cholinesterase Inhibitors: The sample comprised patients evaluated from June, 2009 until October, 2011.During this period, 71 patients were evaluated at baseline and after 3 month-treatment. Donepezil, rivastigmine or galantamine were prescribed to the patients according to the clinicians' preferences. The target dosages considered for treatment effect evaluation were 5 to 10 mg for donepezil, 16 to 24 mg for galantamine and 6 to 12 mg for rivastigmine. The first investigator (LFJRM) did not have any influence on the prescription.
Arm/Group | Patients Taking Cholinesterase Inhibitors
Number analyzed (Participants) | 71
Age, Customized [Count of Participants; unit: Participants]
  ≤ 69 years old | 12
  70-79 years old | 36
  ≥ 80 years old | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 71

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Response After Three Months of Treatment With ChEI in Mild and Moderate Alzheimer's Disease
Description: Patients presented mild or moderate dementia according to the Clinical Dementia Rating (CDR). None of the individuals had been treated with Cholinesterase inhibitors (ChEI) or memantine before study entry. Donepezil, galantamine or rivastigmine were prescribed to the patients according to the clinicians' preferences. All participants were evaluated by one board certified geriatrician (LFJRM) at baseline and after 3 months of treatment, as part of an ongoing 12-month responder analysis study of ChEI in Alzheimer's Disease. The main domain examined and the evaluation tools was cognition and Mini-Mental State Examination- MMSE, respectively. MMSE scores range from 0 to 30, while the greater value is associated with a better cognition state. An increase of 2 or more points in MMSE was considered as response.
Time Frame: three months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CDR 1 Patients Taking Cholinesterase Inhibitors; CDR 2 Patients Taking Cholinesterase Inhibitors: The sample comprised patients evaluated from June, 2009 until October, 2011.During this period, 71 patients were evaluated at baseline and after 3 month-treatment. Donepezil, rivastigmine or galantamine were prescribed to the patients according to the clinicians' preferences. The target dosages considered for treatment effect evaluation were 5 to 10 mg for donepezil, 16 to 24 mg for galantamine and 6 to 12 mg for rivastigmine. The first investigator (LFJRM) did not have any influence on the prescription.
Arm/Group | CDR 1 Patients Taking Cholinesterase Inhibitors | CDR 2 Patients Taking Cholinesterase Inhibitors
Number analyzed (Participants) | 43 | 28
units on a scale
  MMSE- baseline | 19 (4.3) | 11.3 (2.4)
  MMSE - 3 months | 18.9 (4.5) | 11.5 (2.8)

2. Secondary Outcome: Independence for Daily Activities Response After Three Months of Treatment With ChEI in Mild and Moderate Alzheimer's Disease
Description: Patients presented mild or moderate dementia according to the Clinical Dementia Rating (CDR). None of the individuals had been treated with Cholinesterase inhibitors (ChEI) or memantine before study entry. Donepezil, galantamine or rivastigmine were prescribed to the patients according to the clinicians' preferences. All participants were evaluated by one board certified geriatrician (LFJRM) at baseline and after 3 months of treatment, as part of an ongoing 12-month responder analysis study of ChEI in AD. The secondary domain examined was independence for daily activities and the evaluation tools used was the brazilian version of the Pfeffer Functional Activities Questionnaire (PFAQ). PFAQ scale range from 0 to 30 points and the greater value is associated with a greater dependence in daily activities.
Time Frame: three months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CDR 1 Patients Taking Cholinesterase Inhibitors | CDR 2 Patients Taking Cholinesterase Inhibitors
Number analyzed (Participants) | 43 | 28
units on a scale
  PFAQ - baseline | 14.9 (8.8) | 26.9 (4.1)
  PFAQ - 3 months | 16.2 (8.8) | 27.1 (3.5)

ADVERSE EVENTS:
Time Frame: 3 months.
Arm/Group | CDR1 Patients Taking Cholinesterase Inhibitors | CDR2 Patients Taking Cholinesterase Inhibitors
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/23
Other Adverse Events (participants affected / at risk) | 0/48 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No